CLINICAL TRIAL: NCT00302770
Title: Efficacy of Quetiapine in Generalised Social Anxiety Disorder, a Double-blind, Placebo-controlled Study
Brief Title: Efficacy of Quetiapine in Generalised Social Anxiety Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated due to poor enrollment
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1449C00008
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Social Anxiety Disorder
Keywords: Patients with SAD
MeSH Terms: conditions — Phobia, Social | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: quetiapine

SUMMARY:
This trial will explore the efficacy of quetiapine in Social Anxiety Disorder, generalized type. The following elements of response will be tested: number of responders to treatment, time to response, effect size as measured with the LSAS

ELIGIBILITY:
Inclusion Criteria:

* Written Confirmed Consent,
* All patients meet the DSM IV criteria for generalized social anxiety disorder,
* A score ≥ 60 on the LSAS,
* male and female aged between 18 and 65 years

Exclusion Criteria:

* Presence of any primary axis I diagnosis other than social anxiety disorder according to DSM-IV,
* alcohol and/or substance abuse according to DSM-IV criteria within the last 12 months,
* any personality disorder as the primary diagnosis, with the exception of avoidant personality disorder,
* patients at risk of suicide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change on Lebowitz Social Anxiety Scale (LSAS) from baseline to endpoint

SECONDARY OUTCOMES:
Number of responders, time to onset of response of sustained response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Netherlands Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Utrecht, Netherlands